CLINICAL TRIAL: NCT03703661
Title: Can a Low Cost, Simple Needle-Aspirated Compression Dressing Reduce Surgical Site Infection Rates of Primarily Closed Ileostomy and Colostomy Reversal Wounds?
Brief Title: Needle-Aspirated Compression Dressing Following Ostomy Reversal
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Sang Won Lee, Professor of Clinical Surgery, Chief, Division of Colorectal Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00812
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Colostomy Stoma; Ileostomy - Stoma; Surgical Site Infection; Wound Complication
Keywords: negative pressure wound therapy
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): primary closure with gauze and adhesive/occlusive dressing
  Interventions: Procedure: Control
- Negative Pressure (Experimental): primary closure with gauze and adhesive/occlusive dressing under negative pressure
  Interventions: Procedure: Needle-Aspirated Negative Pressure Dressing

INTERVENTIONS:
Procedure: Needle-Aspirated Negative Pressure Dressing — dressing consisting of Needle-Aspirated Negative Pressure dressing with gauze and adhesive/occlusive dressing, placed over wound after primary closure
  Arms: Negative Pressure
Procedure: Control — dressing consisting of gauze and adhesive/occlusive dressing, placed over wound after primary closure
  Arms: Control

SUMMARY:
Negative pressure wound dressings have been studied and shown to have applications in decreasing rates of surgical wound infections. This study studies the effect of a low cost needle-aspirated negative pressure compression dressing on rates of wound infection at prior ostomy site in patients undergoing ostomy reversal surgery.

DETAILED DESCRIPTION:
Negative Pressure Wound Therapy (NPWT) will be studied in colorectal surgery patients undergoing ostomy reversal surgery. The immediate goal is to compare primary wound closure against primary closure with needle-aspirated compression dressing, and determine if risk of potential ostomy site wound infections is decreased. The investigators would also like to evaluate if this compression dressing can increase prevalence of complete wound closure by 12 weeks (last planned clinic visit). NPWT using a continuous suction device was shown to decrease surgical site infection (SSI) at ostomy reversal sites undergoing primary closure. There is a lack of published literature studying NPWT dressings without an associated suction device. The investigators will be using a low-cost simple needle-aspirated suction technique to provide negative pressure under a tegaderm/gauze dressing, at the time of placement. Patients will be consented and randomized into a negative pressure group, or a control group consisting of the same dressing under normal pressure. All adult patients undergoing ostomy reversal surgery who consent to the study will be included. Exclusion criteria include prior recurrent skin infections, prior stoma-site infection, or large parastomal hernia. Patients in the negative pressure group will have the pressure under the dressing measured immediately prior to removal on post-operative day 2.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* presence of a loop or end colostomy or ileostomy
* consenting to study and to ostomy reversal

Exclusion Criteria:

* altered mental status or patients unable to sign the informed consent form
* vulnerable patient populations such as prison and ward patients
* patients who are discovered before or during surgery as unable to undergo placement of compression dressing will be excluded.
* Patients with visible protrusion/evidence of large parastomal hernia
* history of recurrent skin & soft tissue infections
* history of previous stoma site infection or complications
* patients with extensive comorbidities (such as cancer involving stoma site, uncontrolled diabetes, etc), Crohn's patients and abdominal wall fistula patients
* patients in who primary closure of wound is deemed inappropriate by the operating surgeon, requiring a different method of stoma site wound management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-08-27 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 30 days post procedure
  Surgical Site Infection

SECONDARY OUTCOMES:
Rate of Wound Closure | 3 weeks post procedure and 12 weeks post procedure
  rate of wound closure at 3 weeks post procedure and 12 weeks post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sang W Lee, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available outside the study group.